CLINICAL TRIAL: NCT01433549
Title: Effect of Recovery Periods on Ocular Comfort During Daily Lens Wear
Brief Title: Lens Wear Schedules and End-of-Day Comfort
Acronym: INVERMERE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Collaborators: University of Waterloo (Other)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: P-373-C-104
Record Dates: First submitted 2011-09-12; First posted 2011-09-14 (Estimated); Results first posted 2013-04-30 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lotrafilcon B / Senofilcon A (Other): Lotrafilcon B worn first, with senofilcon A worn second, as randomized. Each product was worn bilaterally in 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes, over the course of a 12-hour day, for a total of 4 cycles (days).
  Interventions: Device: Lotrafilcon B; Device: Senofilcon A
- Senofilcon A / Lotrafilcon B (Other): Senofilcon A worn first, with lotrafilcon B worn second, as randomized. Each product was worn bilaterally in 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes, over the course of a 12-hour day, for a total of 4 cycles (days).
  Interventions: Device: Lotrafilcon B; Device: Senofilcon A

INTERVENTIONS:
Device: Lotrafilcon B — Commercially marketed, silicone hydrogel, single-vision contact lens FDA-approved for daily wear and extended (overnight) wear up to 6 nights.
  Other Names: AIR OPTIX® AQUA
Device: Senofilcon A — Commercially marketed, silicone hydrogel, single-vision contact lens FDA-approved for daily wear and extended (overnight) wear up to 6 nights.
  Other Names: ACUVUE® OASYS®

SUMMARY:
The purpose of this study was to assess the impact of lens-free (recovery) intervals of varying lengths on end-of-day comfort and tear film changes with daily contact lens wear.

DETAILED DESCRIPTION:
This study was conducted in a cross-over design with two phases. Each phase consisted of four cycles approximately 12 hours in length. During each cycle, contact lenses were worn for 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes. A new pair of contact lenses was dispensed for each 2-hour interval of lens wear. A 12-hour lens-free wear period preceded each phase.

ELIGIBILITY:
Inclusion Criteria:

* Is at least 17 years of age and has full legal capacity to volunteer.
* Is willing and able to follow instructions and maintain the appointment schedule.
* Has had an ocular examination in the last two years.
* Is an adapted soft contact lens wearer.
* Experiences a decrease in ocular comfort through a lens-wearing day.
* Has a current pair of spectacles.
* Has a distance contact lens prescription of +6.00 diopters to -10.00 diopters and an acceptable fit with the study lenses.
* Has astigmatism less than or equal to -1.00 DC.
* Achieves visual acuity of 6/9 or better with the study lenses and with habitual spectacles.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Has any ocular disease.
* Has a systemic condition that may affect a study outcome variable.
* Is using any systemic or topical medications that may affect ocular health.
* Has known sensitivity to the diagnostic pharmaceuticals to be used in the study.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom FAAO, Director, Principal Investigator — Centre for Contact Lens Research, School of Optometry, University of Waterloo
Locations (1):
- University of Waterloo Centre for Contact Lens Research, Waterloo, Ontario, Canada

REFERENCES:
- [Derived] Stahl U, Keir NJ, Landers A, Jones LW. Effect of Short Recovery Periods on Ocular Comfort During Daily Lens Wear. Optom Vis Sci. 2016 Aug;93(8):861-71. doi: 10.1097/OPX.0000000000000912. PMID 27362613

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from one study center located in Canada.
Pre-assignment Details: Of the 44 participants enrolled, 16 were exited from the study prior to randomization (screen failures). Three subjects were randomized/fitted with lenses but discontinued prior to product dispense. This reporting group includes all participants enrolled and dispensed product. A 12-hour lens-free wear period preceded each phase.
Period: Phase 1: First Study Product
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Phase 2: Second Study Product
Arm/Group | Lotrafilcon B / Senofilcon A | Senofilcon A / Lotrafilcon B
Started | 12 | 13
Completed | 12 | 12
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all participants enrolled and dispensed product.
Groups:
- Overall: Lotrafilcon B and Senofilcon A worn in cross-over fashion as randomized. Each product was worn bilaterally in 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes, over the course of a 12-hour day, for a total of 4 cycles (days).
Arm/Group | Overall
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years] | 25 [19 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 10
Region of Enrollment [Number; unit: participants]
  Canada | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean End-of-Day Comfort
Description: As assessed by the participant using a visual analog scale ranging from 0 (extremely uncomfortable) to 100 (very comfortable and fresh) at the end of each 12-hour (approximate) cycle. During each cycle, contact lenses were worn for 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes. A new pair of contact lenses was dispensed for each 2-hour interval of lens wear.
Time Frame: Hour 12
Population: All participants who participated in both phases of the study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Lotrafilcon B: Lotrafilcon B worn worn bilaterally in 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes, over the course of a 12-hour day, for a total of 4 cycles (days).
- Senofilcon A: Senofilcon A worn bilaterally in 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes, over the course of a 12-hour day, for a total of 4 cycles (days).
Arm/Group | Lotrafilcon B | Senofilcon A
Number analyzed (Participants) | 25 | 25
Units on a scale
  Six 2-hr wear intervals/0-min recovery intervals | 48.9 (17.8) | 56.0 (15.9)
  Five 2-hr wear intervals/30-min recovery intervals | 51.4 (17.6) | 53.7 (15.9)
  Four 2-hr wear intervals/60-min recovery intervals | 56.0 (19.8) | 58.8 (13.9)
  Four 2-hr wear intervals/80-min recovery intervals | 51.5 (13.1) | 58.8 (18.0)

2. Secondary Outcome: Mean Non-Invasive Tear Film Break-Up Time (NITBUT)
Description: As assessed by the investigator using a corneal topographer. NITBUT was assessed at the end of each 12-hour (approximate) cycle. During each cycle, contact lenses were worn for 2-hour intervals, separated by lens-free (recovery) intervals of either 0, 30, 60, or 80 minutes. A new pair of contact lenses was dispensed for each 2-hour interval of lens wear. A longer tear film break-up time indicates a more stable tear film and may lead to a more comfortable lens-wearing experience.
Time Frame: Hour 12
Population: All participants who participated in both phases of the study.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Lotrafilcon B | Senofilcon A
Number analyzed (Participants) | 25 | 25
Seconds
  Six 2-hr wear intervals/0-min recovery intervals | 4.6 (1.9) | 4.3 (1.2)
  Five 2-hr wear intervals/30-min recovery intervals | 5.3 (2.2) | 4.7 (2.4)
  Four 2-hr wear intervals/60-min recovery intervals | 4.4 (2.2) | 4.4 (2.4)
  Four 2-hr wear intervals/80-min recovery intervals | 4.9 (2.6) | 4.8 (2.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (6 months). The safety population is defined as all subjects exposed to product and includes three subjects randomized/fitted with lenses but discontinued prior to product dispense.
Description: The lens wear regimen in this study was not typical. The study protocol required multiple lens insertions and removals within a wear day, which may have negatively impacted ocular surface characteristics in some subjects.
Arm/Group | Lotrafilcon B | Senofilcon A
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28
Other Adverse Events (participants affected / at risk) | 7/28 | 0/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lotrafilcon B (N=28) | Senofilcon A (N=28)
Redness with Indentation (Eye disorders) | 5 | 0
Staining (Eye disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.